CLINICAL TRIAL: NCT05010460
Title: Roxadustat Reduces the Incidence of Acute Kidney Injury After Coronary Artery Bypass Grafting: a Multicenter, Randomized, Double-blind, Placebo-controlled Study
Brief Title: Study of Roxadustat for Reducing the Incidence of Acute Kidney Injury After Coronary Artery Bypass Grafting
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow enrollment and inability to reach the planned sample size within the expected timeframe
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ROXAKI
Record Dates: First submitted 2021-08-07; First posted 2021-08-18 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Bypass
Keywords: acute kidney injury; coronary artery bypass; Roxadustat
MeSH Terms: conditions — Acute Kidney Injury | interventions — roxadustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Roxadustat (Experimental): Roxadustat
  Interventions: Drug: Roxadustat
- placebo (Placebo Comparator): Placebo has the same appearance with the experimental drug (Roxadustat).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Roxadustat — orally 100mg every other day for 5-8 days prior to CABG
  Other Names: Evrenzo
  Arms: Roxadustat
Drug: Placebo — orally 100mg every other day for 5-8 days prior to CABG
  Arms: placebo

SUMMARY:
Acute kidney injury is a frequent complication after coronary artery bypass grafting (CABG). Roxadustat is a prolyl hydroxylase inhibitor (PHI) which can stabilize hypoxia-inducible factor (HIF) and improve the hypoxic tolerance of tissues. Roxadustat has shown effect in reducing acute kidney injury in animal studies.

This study aims to evaluate the efficacy of administration of Roxadustat before surgery in the prevention of acute kidney injury after CABG.

DETAILED DESCRIPTION:
Acute kidney injury is a frequent complication after coronary artery bypass grafting (CABG), with a incidence of 28-38%. Renal ischemia-reperfusion injury is the main mechanism for acute kidney injury after CABG.

Roxadustat is a kind of prolyl hydroxylase inhibitor (PHI) which can stabilize hypoxia-inducible factor (HIF) and improve the hypoxic tolerance of tissues. Roxadustat has shown effect in reducing acute kidney injury in animal studies.

This study aims to evaluate the efficacy of administration of Roxadustat (before surgery) in the prevention of acute kidney injury after CABG. This is a multicenter, randomized, double-blind, placebo-controlled study.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* non-emergent CABG and planned cardiopulmonary bypass (CPB)
* eGFR>15ml/min/1.73m2

Exclusion Criteria:

* pregnancy or breast feeding
* malignancy
* severe liver dysfunction
* acute kidney injury before randomization
* uncontrolled hypertension

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
acute kidney injury | 0-48 hours after surgery
  elevation of serum creatinine ≥0.3mg/dl（26.5μmol/L）or ≥ 1.5 times baseline levels within 48 hours post surgery

SECONDARY OUTCOMES:
classification of acute kidney injury | 0-3 days after surgery
  classification of of acute kidney injury based on AKIN criteria
renal function | 0-3 days after surgery
  creatinine, urea, Cystatin-C after surgery
new biomarkers of renal injury | immediately after surgery and the first morning after surgery
  serum and urine NGAL，urine TIMP2*IGFBP7
Cardiac Troponin Subunit I (cTnI) | 0-3 days after surgery
  peak plasma concentration of cTnI and area under curve (AUC) of cTnI
brain natriuretic peptide (BNP) or N-terminal pro-BNP (NT-proBNP) | 0-3 days after surgery
  plasma concentration of BNP
death | through study completion, an average of one month
  death during hospitalization
length of hospital stay and ICU stay | through study completion, an average of one month
  length of hospital stay and ICU stay
Blood infusion | 0-3 days after surgery
  amount of Red blood cells infusion after surgery
adverse events | through study completion, an average of one month
  adverse events and severe adverse events during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Yan Qin, Doctor, Principal Investigator — Peking Union Medical College Hospital; Qi Miao, Doctor, Principal Investigator — Peking Union Medical College Hospital
Locations (2):
- China (2):
  - Beijing Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Yes
qualified researchers can request access to anonymized individual patient-level data by contacting principle investigator of this study, but this does not mean all requests will be shared by the investigators.
Supporting Information: Study Protocol, SAP
Time Frame: 1 year after the end of this study
Access Criteria: please contact the investigators through email in the time frame

REFERENCES:
- [Background] Chertow GM, Burdick E, Honour M, Bonventre JV, Bates DW. Acute kidney injury, mortality, length of stay, and costs in hospitalized patients. J Am Soc Nephrol. 2005 Nov;16(11):3365-70. doi: 10.1681/ASN.2004090740. Epub 2005 Sep 21. PMID 16177006
- [Background] Hill P, Shukla D, Tran MG, Aragones J, Cook HT, Carmeliet P, Maxwell PH. Inhibition of hypoxia inducible factor hydroxylases protects against renal ischemia-reperfusion injury. J Am Soc Nephrol. 2008 Jan;19(1):39-46. doi: 10.1681/ASN.2006090998. PMID 18178798
- [Background] Shu S, Wang Y, Zheng M, Liu Z, Cai J, Tang C, Dong Z. Hypoxia and Hypoxia-Inducible Factors in Kidney Injury and Repair. Cells. 2019 Feb 28;8(3):207. doi: 10.3390/cells8030207. PMID 30823476
- [Background] Kapitsinou PP, Jaffe J, Michael M, Swan CE, Duffy KJ, Erickson-Miller CL, Haase VH. Preischemic targeting of HIF prolyl hydroxylation inhibits fibrosis associated with acute kidney injury. Am J Physiol Renal Physiol. 2012 May 1;302(9):F1172-9. doi: 10.1152/ajprenal.00667.2011. Epub 2012 Jan 18. PMID 22262480
- [Background] Chen N, Hao C, Peng X, Lin H, Yin A, Hao L, Tao Y, Liang X, Liu Z, Xing C, Chen J, Luo L, Zuo L, Liao Y, Liu BC, Leong R, Wang C, Liu C, Neff T, Szczech L, Yu KP. Roxadustat for Anemia in Patients with Kidney Disease Not Receiving Dialysis. N Engl J Med. 2019 Sep 12;381(11):1001-1010. doi: 10.1056/NEJMoa1813599. Epub 2019 Jul 24. PMID 31340089